CLINICAL TRIAL: NCT05683379
Title: Anti-AAV8 Antibody Assessment Study of Males With Duchenne Muscular Dystrophy Aged 0 to <25 Years
Brief Title: AFFINITY BEYOND: Anti-AAV8 Antibody Assessment Study of Males With DMD
Status: Recruiting | Type: Observational
Sponsor: REGENXBIO Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RGX-202-0101
Record Dates: First submitted 2023-01-04; First posted 2023-01-13 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: DMD; Duchenne Muscular Dystrophy; Duchenne
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

INTERVENTIONS:
Diagnostic Test: AAV8 DetectCDx — An in vitro diagnostic assay to detect antibodies to AAV8 in human serum specimens.

SUMMARY:
This is an observational screening study to evaluate the prevalence of anti-adeno-associated serotype 8 (AAV8) antibodies in participants with Duchenne muscular dystrophy (DMD).

DETAILED DESCRIPTION:
This is an observational screening study to evaluate the prevalence of anti-adeno-associated serotype 8 (AAV8) antibodies in participants with Duchenne muscular dystrophy (DMD). Information collected in this study may be used to identify potential participants for DMD investigational gene therapy clinical trials.

This study consists of:

* A phone/video interview or at an in-clinic visit to provide e-consent and medical history
* A single home health visit or subsequent in-clinic visit to collect blood sample for antibody testing
* A phone/video call for communication of AAV8 antibody test results

ELIGIBILITY:
Inclusion Criteria:

* Males at least 0 to <25 years of age
* Diagnosis of DMD
* Provision of signed and dated informed consent form (ICF) and assent as required per local regulations or requirements

Exclusion Criteria:

* Prior participation in a gene therapy trial OR recipient of a gene therapy drug
* Other inclusion/exclusion criteria apply

Ages: 0 Years to 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Primary care clinic, Musculoskeletal care, Neuromusculoskeletal care
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Prevalence of anti-AAV8 antibodies in patients with DMD | 90 days
  * To evaluate the prevalence of AAV8 antibodies in patients with DMD
  * To identify participants who may be eligible for investigational gene therapy clinical trials in males with DMD

CONTACTS AND LOCATIONS:
Locations (1):
- Rare Disease Research, Atlanta, Georgia, United States